CLINICAL TRIAL: NCT06574100
Title: Relative Bioavailability of Two Orally Administered CBD Formulations in Healthy Male Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: University of Regina (Other)
Responsible Party: Principal Investigator, Jane Alcorn, Dean and Professor at the College of Pharmacy and Nutrition, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NFL-CBD-02; Bio-4317 (Other: University of Saskatchewan Research Ethics Board); 286992 (Other: Health Canada NOL control #)
Record Dates: First submitted 2024-06-28; First posted 2024-08-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: We plan this study as a single-site (potentially multi-site), randomized, two-arm study, with one arm being a two-sequence crossover, single buccal, or oral dose in fasted healthy male adults, and the second arm being a two-sequence cross-over, single high oral dose PK study in fasted vs fed-state healthy male adults. Participants will be randomized into four groups (n = 16 in Arm 1, 8 per group (2 groups), all males; n = 4 in Arm 2, 2 per group (2 groups) all males) (ages 18 - 35) based on which formulation each group will receive. Individuals in study arm 1 will complete the study in the fasted state (10 hours of fasting). Individuals in study arm 2 will follow the fed-state protocol as outlined by the United States FDA's bioequivalent studies guideline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Single Oral Dose Administration of 250mg Buccally or 1000 mg Orally of two CBD formulations (Active Comparator): participants receiving the buccal formulation will be required to receive 10 strips by the cheeks, they will be instructed to only swallow at maximum once every 2 mins for the first 5 mins. This is to minimize the amount of CBD that will be carried into the GIT. This buccal administration group will receive 2 strips at a time, one on each cheek side, following 5 mins of dissolving, patients will receive 100mL of water to swish the residue in their mouths and swallow, then receive another pair of strips to repeat the process for a total of 5 times over the course of 30 minutes (i.e., 10 strips total). The group receiving the 1000mg oral CBD extract will mimic the buccal group in that they will receive that dose over the course of 30 minutes in 5 parts, 200mg per part, and will drink 100mL of water to accompany its administration
  Interventions: Drug: Cannabidiol
- Single Oral Dose Administration of 3000mg CBD Extract in Fed vs Fasting (Active Comparator): In the fasting group, participants will be asked to fast overnight (at least 10 hours fast) but are allowed to drink water.In the fed state group, participants will start their meal 30 minutes prior to receiving the dose. The meal will consist of high caloric (800-1000 Cal), high fat (~50% of total calories), with protein, and carbohydrates (~150 kcal, and ~250 kcal, respectively) content. No food will be administered 4 hours after the dose, and no water will be given 1 hour prior to dose administration and 1 hour after administration. The dose will be given however with a total of 235 mL of water.
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Patients in the first arm cross-over will receive either a single bolus dose of 250mg buccally administered or 1000mg CBD powder and cross over to vice-versa after 21 days.
  Other Names: One formulation will be a powder the other will be buccal strips
  Arms: Single Oral Dose Administration of 250mg Buccally or 1000 mg Orally of two CBD formulations
Drug: Cannabidiol — Patients will be randomised to receive 3000mg oral CBD fasting or Fed, they will the cross over to the other group 21 days following the first administration.
  Arms: Single Oral Dose Administration of 3000mg CBD Extract in Fed vs Fasting

SUMMARY:
This project is aimed at understanding whether a new fast-dissolving cheek-administered cannabidiol strip will be absorbed better into the body than cannabidiol powder. The results of this study will help guide dosage formulation choices as well as dosing regimens in NFL athletes for concussion management.

DETAILED DESCRIPTION:
Cannabis formulations are typically administered by the oral route of administration. This route represents the most common administration route for most pharmaceuticals due to the ease of administration and convenience. Inhalational products are not acceptable for the sport's athlete population due to potential damage to lung tissues. Topical products do not have adequate bioavailability to meet our therapeutic objectives. Our PK studies, then, need to employ the same dosage form and route of administration we expect to use in future clinical efficacy trials.

Given the low bioavailability expected with CBD oral formulations, we wish to assess two different formulations and the relative extent of CBD absorption. Our future planned CBD intervention studies in athletes will require use of larger doses of CBD. The formulation with the larger bioavailability will help to reduce the overall size of the dose utilized and therefore reduce the amount of product exposure in our clinical intervention studies. This will increase the likelihood that a Cannabis company can supply the necessary amount of product and reduce the overall cost associated with the studies. Generally speaking, based on current literature published around CBD administration for therapeutic application, higher doses of CBD (i.e., 50mg/kg/d) were found to correlate to more positive outcomes than lower doses (i.e., 1mg/kg/d). Assuming an average weight of 70 kg, a 1000 mg dose would be around 14.29 mg/kg, and a 3000 mg dose around 42.86 mg/kg. This will allow us to investigate the pharmacokinetics of CBD on both ends of the hypothetical efficacy trend. Studies have examined single orally administered doses up to 6000 mg with no serious adverse effects reported.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 35 years old
2. Clinical labs within the stated normal range of the Royal University Hospital Test Centre, or values outside the stated normal range that are not of clinical significance as determined by the qualified investigator.
3. No clinically significant disease on medical history or clinically significant findings on physical examination including vital signs as determined by the qualified investigator.
4. Ability to stay in the clinic trial unit for 13 hours on the day of each single oral dose.
5. Ability to return for blood draws in the subsequent days.

Exclusion Criteria:

1. History or presence of significant gastrointestinal, liver or kidney disease or any other condition known to interfere with drug pharmacokinetics including bioavailability or increase risk of adverse effects.
2. History or presence of serious cardiovascular disease, such as ischaemic heart disease, arrhythmias, poorly controlled hypertension or severe heart failure
3. Males whose partners are trying to conceive (i.e. male subjects intending to start a family during the study period)
4. Lack of medically acceptable contraception by participants whose female partners have childbearing potential for the duration of the study.
5. Personal or family history of schizophrenia or any other psychotic disorder
6. Current or past drug or alcohol dependence or abuse
7. Use of Cannabis-based therapy within 2 months (Participants who have previously used a Cannabis-based therapy may be included if they have a 2-month period without use of Cannabis-based therapy prior to enrolment in the study)
8. Use of recreational Cannabis within 2 months (Participants who have previously used recreational Cannabis may be included if they have a 2-month period without use of recreational Cannabis prior to enrolment in the study)
9. Use of psychotropic medications with serotonergic activity (e.g. Selective Serotonin Reuptake Inhibitors, Tricyclic Antidepressants, Atypical Neuroleptics) within one week
10. Use of narcotic medications (e.g. Codeine, Morphine, Oxycontin) within one week
11. Use of any other medication known to interact with medicinal Cannabis within one week.
12. Allergy or known intolerance to any of the compounds within the study preparation.
13. Resting heart rate HR < 50 bpm or > 100 bpm or seated blood pressure < 100/60 or higher than 140/90
14. Inability of study participants to attend and complete all study visits
15. Bleeding disorder
16. Known low hematocrit

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-26 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Parameters | 1 week of samples will be collected. 2 week washout. Then another week of samples after cross over
  relative bioavailability (F)
Pharmacokinetic Parameters | 1 week of samples will be collected. 2 week washout. Then another week of samples after cross over
  time to maximum plasma concentration (Tmax)
Pharmacokinetic Parameters | 1 week of samples will be collected. 2 week washout. Then another week of samples after cross over
  maximum plasma concentration (Cmax)
Pharmacokinetic Parameters | 1 week of samples will be collected. 2 week washout. Then another week of samples after cross over
  log-linear terminal phase rate constant (k)
Pharmacokinetic Parameters | 1 week of samples will be collected. 2 week washout. Then another week of samples after cross over
  area under the plasma concentration versus time curve (AUC)
Pharmacokinetic Parameters | 1 week of samples will be collected. 2 week washout. Then another week of samples after cross over
  absorption rate constant (ka)
Pharmacokinetic Parameters | 1 week of samples will be collected. 2 week washout. Then another week of samples after cross over
  apparent clearance (Cl/F)
Pharmacokinetic Parameters | 1 week of samples will be collected. 2 week washout. Then another week of samples after cross over
  apparent volume of distribution (Vd/F)
Pharmacokinetic Parameters | 1 week of samples will be collected. 2 week washout. Then another week of samples after cross over
  half-life

SECONDARY OUTCOMES:
Safety of the drug using the Integrated Addendum to ICH E6(R1) | During the first week of administration and the 4th week of administration
  Safety of the study drug will be determined by measuring blood pressure (mmhg)
Safety of the drug using the Integrated Addendum to ICH E6(R1) | During the first week of administration and the 4th week of administration
  Safety of the study drug will be determined by measuring heart rate (beats/minute)
Safety of the drug using the Integrated Addendum to ICH E6(R1) | During the first week of administration and the 4th week of administration
  Safety will be assessed by reporting of incidence of adverse events for each participant.
Optimal washout periods | 3 weeks
  Measure CBD and it's metabolites over the course of the study to determine what the optimal washout period is for future studies
Tolerability of the drug using the Integrated Addendum to ICH E6(R1) | During the first week of administration and the 4th week of administration
  Tolerability of the study drug will be determined by reporting of incidence of adverse events for each participant.
Compare Fed vs Fast state on oral absorption kinetics | 1 week of samples will be collected. 2 week washout. Then another week of samples after cross over
  half-life
Compare Fed vs Fast state on oral absorption kinetics | 1 week of samples will be collected. 2 week washout. Then another week of samples after cross over
  apparent volume of distribution (Vd/F)
Compare Fed vs Fast state on oral absorption kinetics | 1 week of samples will be collected. 2 week washout. Then another week of samples after cross over
  apparent clearance (Cl/F)
Compare Fed vs Fast state on oral absorption kinetics | 1 week of samples will be collected. 2 week washout. Then another week of samples after cross over
  absorption rate constant (ka)
Compare Fed vs Fast state on oral absorption kinetics | 1 week of samples will be collected. 2 week washout. Then another week of samples after cross over
  area under the plasma concentration versus time curve (AUC)
Compare Fed vs Fast state on oral absorption kinetics | 1 week of samples will be collected. 2 week washout. Then another week of samples after cross over
  log-linear terminal phase rate constant (k)
Compare Fed vs Fast state on oral absorption kinetics | 1 week of samples will be collected. 2 week washout. Then another week of samples after cross over
  maximum plasma concentration (Cmax)
Compare Fed vs Fast state on oral absorption kinetics | 1 week of samples will be collected. 2 week washout. Then another week of samples after cross over
  time to maximum plasma concentration (Tmax)
Compare Fed vs Fast state on oral absorption kinetics | 1 week of samples will be collected. 2 week washout. Then another week of samples after cross over
  relative bioavailability (F)

CONTACTS AND LOCATIONS:
Overall Officials: Payam Dehghani, MD, Principal Investigator — Pasqua Hospital; Jane Alcorn, DVM;PhD, Principal Investigator — University of Saskatchewan; Abdul Salama, PharmD, Study Director — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Undecided